CLINICAL TRIAL: NCT04049968
Title: Using an APP in Post Oral Cancer Surgery to Affect Patients' Needs and Quality of Life.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 105110-E
Record Dates: First submitted 2019-08-04; First posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2016-11

CONDITIONS: Oral Cancer
Keywords: Oral cancer、Post-Operation Needs、Quality of Life、APP
MeSH Terms: conditions — Mouth Neoplasms | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Patients were divided into two two groups. Control group was assessed with traditional routine healthcare and instruction. Experimental group was assessed with a mobile health application.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients in the experimental group were individually assessed by a mobile health application (APP).
  Interventions: Device: Mobile health application (APP)
- Control group (Active Comparator): Patients in the control group were individually assessed by a traditional routine health care and instruction.
  Interventions: Other: Routine health care and instruction

INTERVENTIONS:
Device: Mobile health application (APP) — The mobile health application (APP) was applied to patients with oral cancer.
  Arms: Experimental group
Other: Routine health care and instruction — Traditional routine health care and instruction was applied to patients with oral cancer.
  Arms: Control group

SUMMARY:
This study aimed to explore using an APP in post oral cancer surgery to affect patients' needs and quality of life.

Methods Quasi-experimental Research Design used purposeful sampling from January 1 to December 31 of the Far Eastern Memorial Hospital oral maxillofacial surgery ward and the otolaryngology ward requirement met post-treatment oral cancer patients who agreed to participate. Self-administered structured questionnaires, including basic personal information, cancer needs table short version (CNQ-SF), head and neck cancer quality of life scale (EORTC QLQ-H&N35), were used to collect information. Results were statistically analyzed to understand the distribution of variables and their relationships.

Scientific or Clinical Implication of the Expected Results Using an APP intervention in post-operative patients with oral cancer may be the better way to promote health and enhance one's quality of life.

DETAILED DESCRIPTION:
The malignant tumor has been consecutively ranked as number one of the top ten causes of death over the past 33 years, and the incidence of an increase in oral cancer year by year. The average age of death was 55-57. With this average age compared to other cancer patients under 10 years of early life, it's necessary to care about the burden of disease from oral cancer. The main treatment of oral cancer is surgery and a combination of radiotherapy and chemotherapy. Patients often got severe treatment complications with varying degrees of physical functions and uncertainty due to poor cognition or less clarification in a complex course of treatment that affects medical decisions in the illness process. Both domestic and foreign research show that the majority of oral cancer patients expressed the need for and attention to health information. "Treatment information" was the most needed and important. When information needs are met, it can effectively reduce the anxiety and unease of unknown events. Relevant domestic and foreign research do not provide accessibility and convenience of health education for post-operative patients with oral cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed with oral cancer and were the first-time receiving oral cancer surgery within 1 week.
* Conscious and able o communicate
* Patients agreed to participate in this study and had a smart phone.

Exclusion Criteria:

* Patients without oral cancer
* Patients with oral cancer but had received oral cancer surgery before 1 week or more.
* Unconscious or unable to answer questions from questionnaire or APP
* Patients with cognitive impairment, dementia o intellectual disability.

Ages: 48 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Changes of the subjects' quality of life | 3 month
  The Quality of Life scale (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, Core Module [EORTC QLQ-C30] and Head and Neck Module [QLQ-H&N35], or EORTC QLQ-H&N35) was used to represent patients' satisfaction with quality of life. The EORTC QLQ-H&N35 is a 30-item self-administered global health and quality of life questionnaire with 5 scales, including physical, role, cognitive, emotional and social functioning. In addition, the measuring items included the pain, swallowing, speech, taste/smell, eating, dry mouth, coughing, opening mouth and social contact and sexuality.
Changes of the subjects' physiological needs | 3 month
  Care Needs Scale (the short-form Cancer Needs Questionnaire, CNQ-SF) was used to measure baseline postoperative care needs, with score 0 meaning no care need and score 100 meaning highest care need. CNQ-SF is a 32-item self-administered questionnaire to evaluate five domains of patient needs, including psychological, health information, physical and daily living, patient care and support, and interpersonal communication needs.

SECONDARY OUTCOMES:
Changes of the subjects' response to health IT | 3 month
  Science and Technology Acceptance Model scale was applied to evaluate patients' response to health IT. The scale measures subjects' intention, perceived usefulness, and perceived ease of use. Effectiveness is determined by a panel of experts, including nursing experts, nursing information experts and medical information experts.

CONTACTS AND LOCATIONS:
Overall Officials: Lee-Chen Chen, Principal Investigator — Far Eastern Memorial Hospital

IPD SHARING:
Plan to Share IPD: No
The data is currently under analysis.

REFERENCES:
- [Derived] Wang TF, Huang RC, Yang SC, Chou C, Chen LC. Evaluating the Effects of a Mobile Health App on Reducing Patient Care Needs and Improving Quality of Life After Oral Cancer Surgery: Quasiexperimental Study. JMIR Mhealth Uhealth. 2020 Jul 27;8(7):e18132. doi: 10.2196/18132. PMID 32716303